CLINICAL TRIAL: NCT07277322
Title: Master Protocol for A Phase 1b/2 Study of Neoadjuvant Immunotherapy in Microsatellite Stable (MSS) Colorectal Cancer (CRC) Subjects With Resectable Liver Metastases
Brief Title: Neoadjuvant Dupilumab and Toripalimab in MSS CRC Subjects With Resectable Liver Metastases
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dan Feng (Other)
Collaborators: Coherus Oncology, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Dan Feng, Assistant Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STUDY-25-01112; PRMC-25-088 IIT (Other: Icahn School of Medicine at Mount Sinai)
Record Dates: First submitted 2025-12-02; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Colorectal Cancer; Liver Metastases
Keywords: Colorectal cancer; Liver metastases; Neoadjuvant immunotherapy; Dupilumab; Toripalimab; microsatellite stable
MeSH Terms: conditions — Colorectal Neoplasms | interventions — dupilumab; toripalimab

STUDY DESIGN:
Intervention Model Description: Safety run-in phase of at most 6 subjects, guided by a 3+3 design. Phase 2: After enrolling 12 patients in the first stage, the trial will be terminated if no radiological responses are observed. If at least one response is observed, 9 additional patients will be enrolled for a total of 21. If 3 or more radiological responses are observed in the full cohort, the null hypothesis will be rejected and the treatment considered for further study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dupilumab and toripalimab (Experimental): Participants will receive the combination of Dupilumab and Toripalimab
  Interventions: Drug: Dupilumab; Drug: Toripalimab

INTERVENTIONS:
Drug: Dupilumab — Dupilumab is commercially sourced, and provided as 300mg pre-filled syringes, though packaging may vary. Dupilumab 600mg SC on Day 1 and 300mg SC on Day 15 (+/-2 days).
Drug: Toripalimab — Toripalimab will be supplied as a liquid in sterile, single-use vials that will display the product lot number on the label. Each vial contains 240 mg/6 mL (40 mg/mL) solution. Toripalimab 240mg IV over 60 minutes or longer on Day 1 before planned surgery.

SUMMARY:
This Phase 1b/2 trial will evaluate the safety and efficacy of neoadjuvant immunotherapy in microsatellite stable (MSS) colorectal cancer (CRC) subjects with resectable liver metastases.

DETAILED DESCRIPTION:
This is a Phase 1b/2 study of neoadjuvant dupilumab and toripalimab in MSS CRC subjects with resectable liver metastases. The primary objective of Phase 1b is to determine the safety of neoadjuvant immunotherapy in MSS CRC subjects with resectable liver metastases. The primary objective of Phase 2 is to determine the efficacy of immunotherapy in MSS CRC subjects with resectable liver metastases as measured by the percentage of subjects achieving a major pathological response (MPR). Eligible subjects will receive dupilumab (600mg on Day 1 and 300mg on D15 ±2 days) and toripalimab 240mg on Day 1 before planned surgery. Dupilumab is administered as a subcutaneous injection. Toripalimab is administered intravenously over 60 minutes or longer. Based on clinical signal in the current cohort and new findings in animal models, additional cohorts will be added to test different immunotherapy combinations in the same patient population with the same endpoints and statistical method in the future.

ELIGIBILITY:
INCLUSION CRITERIA:

Histological diagnosis of non-MSI-H/pMMR CRC

• Subjects who have biology-proven non-MSI-H/pMMR CRC and with radiographic findings suggestive of liver metastases may be eligible.

Resectable liver metastases including:

* synchronous liver metastases (present at the time of diagnosis of MSS CRC) and treatment-naïve
* metachronous liver metastasis (developed after resection of the primary tumor) without prior adjuvant chemotherapy
* metachronous liver metastasis (developed after resection of the primary tumor) with adjuvant chemotherapy completed greater than 3 months from the time of consent.

Surgical candidate for resection

Age ≥ 18 years. Rationale: Because no dosing or adverse event data are currently available on the use of dupilumab in combination with toripalimab in subjects <18 years of age, children are excluded from this study.

ECOG Performance Status 0-1 (Karnofsky ≥60%,)

• Subjects with performance status >1 carrying long-term disability (such as cerebral palsy) where the disability is not acute nor progressive, and unlikely to significantly affect their response to therapy may be enrolled at the investigator's discretion

Women of child-bearing potential (WOCBP) and men must agree to use adequate contraception upon study entry, for the duration of study participation, and for 3 months following completion of therapy.

* A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

  * Has not undergone a hysterectomy or bilateral oophorectomy; or
  * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).

Ability to understand and the willingness to sign a written informed consent. Legally authorized representatives may sign and give informed consent on behalf of study participants.

Adequate organ and marrow function as defined:

* Hematologic

  o Absolute neutrophil count (ANC) ≥1,000 /mcL
  * Platelets ≥75,000 /mcL
  * Hemoglobin ≥8 g/dL
* Renal* o Serum creatinine ≤1.5 X upper limit of normal (ULN) OR Measured or calculated (Creatinine clearance should be calculated per institutional standard) creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≥45 mL/min for subjects with creatinine levels > 1.5 X institutional ULN
* Hepatic* o Serum total bilirubin ≤ 1.5 X ULN OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN; ≤ 3 X ULN for subjects with liver metastases o AST ≤ 2.5 X ULN OR ≤ 5 X ULN for subjects with liver metastases

  * ALT ≤ 2.5 X ULN OR ≤ 5 X ULN for subjects with liver metastases
  * Albumin >2.5 mg/dL
* Coagulation*

  * International Normalized Ratio (INR) or Prothrombin Time (PT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT is within therapeutic range of intended use of anticoagulants
  * Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PTT is within therapeutic range of intended use of anticoagulants * If laboratory criteria are not met due to what the investigator determines to be a biologic cause (e.g. Gilbert's syndrome causing elevated bilirubin or excessive muscle mass affecting creatinine) or drug-related cause (e.g. elevating in transaminases due to HAART therapy, elevated INR due to anticoagulation) then the lab values will not be used to exclude subject from this trial. This determination will be made by PI.

EXCLUSION CRITERIA:

History of autoimmune disorder with the following exceptions:

* Vitiligo, alopecia, psoriasis or any chronic skin condition that does not require systemic therapy
* Hypothyroidism (e.g. following autoimmune thyroiditis) stable on thyroid replacement
* Celiac disease controlled by diet alone

Treatment, for any reason, with an immunomodulatory drug, within 8 weeks from time of consent.

Prior treatment with dupilumab within the last 8 weeks.

Prior treatment with chemotherapy for MSS CRC or locoregional therapy to the target lesion (that will be biopsied and subsequently resected) within 3 months prior to entering the study.

• Previous therapy for a different cancer (a different primary) is acceptable.

Use of investigational agents for treatment of cancer.

Subjects with extrahepatic metastases that are not amendable to resectable or locoregional therapy, for whom the intent of surgery would not be curative.

Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection requiring antibiotics (exception is a brief (≤10 days) course of antibiotics to be completed before initiation of treatment), symptomatic congestive heart failure, unstable angina pectoris, or psychiatric illness/social situations that would limit compliance with study requirements, as determined the treating investigator.

Pregnant or nursing women due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants.

• Breastfeeding should be discontinued prior to study enrollment.

Has a diagnosis of primary immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.

• Chronic steroids equivalent to ≤ 10mg prednisone are permitted.

Has active autoimmune disease that has required systemic treatment in the past 1 year (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs).

• Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is permitted.

Has a known additional malignancy that is progressing and requires active treatment.

• Exceptions include: basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical or anal cancer, prostate cancer on stable dose of hormonal therapy without rising PSA, and breast cancer treated with curative intent now on hormonal therapy.

Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating Investigator.

HIV positive with detectable viral load, or anyone not on stable anti-viral (HAART) regimen, or with <200 CD4+ T cells/microliter in the peripheral blood. HIV testing is mandatory for patients with no known history of HIV. For such patients, HIV testing will be considered SOC.

Has known active Hepatitis B (e.g., HBV detected by PCR (>200 IU/ml) or known active Hepatitis C (e.g., HCV RNA [qualitative] is detected).

• Subjects who started antiviral therapy >/=14days from baseline are permitted.

History of allogeneic hematopoietic cell transplantation or solid organ transplantation.

Documented allergic or hypersensitivity response to any protein therapeutics (e.g., recombinant proteins, vaccines, intravenous immune globulins, monoclonal antibodies, receptor traps) Principle investigator believes that for one or multiple reasons the subject will be unable to comply with all study visits, or if they believe the trial is not clinically in the best interest of the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2030-12-16 (Estimated); Study Completion 2030-12-16 (Estimated)

PRIMARY OUTCOMES:
Number of dose limiting toxicities (DLTs) | up to 30 days post last administration of study drug dupilumab
  Phase 2: Safety of treatment, defined as the frequency and percentage of DLTs, from start of treatment up to 30 days post the last administration of study drug (dupilumab).

SECONDARY OUTCOMES:
Major pathological response (MPR) | Day of Surgery (day 16-22)
  Major pathological response (MPR), defined as the presence of viable tumor cells in less than 10% of the target lesion.
Time to surgery | up to 22 days
  Time from the initial dose of dupilumab to the time of surgery, measured in days.
Percentage of participants with adverse event | within 90 days following the final dose of dupilumab
  Safety and tolerability defined by the percentage of individuals who experience adverse events (according to NCI CTCAE v5.0) at any point during the neoadjuvant period, or within 90 days following the final dose of dupilumab received, that are attributable to dupilumab and/or toripalimab,
Event free survival (EFS) | Initial treatment to progression of disease, recurrence of tumor following surgery, up to 8 weeks, whichever comes first after first dose of dupilumab,
  Time from initial treatment of dupilumab and toripalimab to progression of disease, recurrence of tumor following surgery, or death from any cause regardless of etiology.
Overall survival (OS) | From treatment initiation until death from any cause, up to 2 years, whichever comes first
  Time, in days, between treatment initiation and when the subject dies from any cause regardless of etiology

CONTACTS AND LOCATIONS:
Overall Officials: Dan Feng, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Thomas Marron, MD, PhD, Study Chair — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
The completed dataset is the sole property of the Sponsor-Investigator's institution and should not be exported to third parties, except for authorized representatives of appropriate Health/Regulatory Authorities, without permission from the Sponsor-investigator and their institution.

REFERENCES:
- [Background] Fakih M, Sandhu J, Wang C, Kim J, Chen YJ, Lai L, Melstrom K, Kaiser A. Evaluation of Comparative Surveillance Strategies of Circulating Tumor DNA, Imaging, and Carcinoembryonic Antigen Levels in Patients With Resected Colorectal Cancer. JAMA Netw Open. 2022 Mar 1;5(3):e221093. doi: 10.1001/jamanetworkopen.2022.1093. PMID 35258578
- [Background] Pellini B, Chaudhuri AA. Circulating Tumor DNA Minimal Residual Disease Detection of Non-Small-Cell Lung Cancer Treated With Curative Intent. J Clin Oncol. 2022 Feb 20;40(6):567-575. doi: 10.1200/JCO.21.01929. Epub 2022 Jan 5. PMID 34985936
- [Background] Brown B. How a hobby farm taught me to set priorities in academia. Nature. 2022 Oct 5. doi: 10.1038/d41586-022-03184-8. Online ahead of print. No abstract available. PMID 36198820
- [Background] Martins F, Sofiya L, Sykiotis GP, Lamine F, Maillard M, Fraga M, Shabafrouz K, Ribi C, Cairoli A, Guex-Crosier Y, Kuntzer T, Michielin O, Peters S, Coukos G, Spertini F, Thompson JA, Obeid M. Adverse effects of immune-checkpoint inhibitors: epidemiology, management and surveillance. Nat Rev Clin Oncol. 2019 Sep;16(9):563-580. doi: 10.1038/s41571-019-0218-0. PMID 31092901
- [Background] Huang AC, Orlowski RJ, Xu X, Mick R, George SM, Yan PK, Manne S, Kraya AA, Wubbenhorst B, Dorfman L, D'Andrea K, Wenz BM, Liu S, Chilukuri L, Kozlov A, Carberry M, Giles L, Kier MW, Quagliarello F, McGettigan S, Kreider K, Annamalai L, Zhao Q, Mogg R, Xu W, Blumenschein WM, Yearley JH, Linette GP, Amaravadi RK, Schuchter LM, Herati RS, Bengsch B, Nathanson KL, Farwell MD, Karakousis GC, Wherry EJ, Mitchell TC. A single dose of neoadjuvant PD-1 blockade predicts clinical outcomes in resectable melanoma. Nat Med. 2019 Mar;25(3):454-461. doi: 10.1038/s41591-019-0357-y. Epub 2019 Feb 25. PMID 30804515
- [Background] Barany F. [News about Crohn disease]. Lakartidningen. 1982 Feb 17;79(7):489-94. No abstract available. Swedish. PMID 7087618
- [Background] Ivanova A, Qaqish BF, Schell MJ. Continuous toxicity monitoring in phase II trials in oncology. Biometrics. 2005 Jun;61(2):540-5. doi: 10.1111/j.1541-0420.2005.00311.x. PMID 16011702
- [Background] Matson V, Fessler J, Bao R, Chongsuwat T, Zha Y, Alegre ML, Luke JJ, Gajewski TF. The commensal microbiome is associated with anti-PD-1 efficacy in metastatic melanoma patients. Science. 2018 Jan 5;359(6371):104-108. doi: 10.1126/science.aao3290. PMID 29302014
- See also: Frank EH. Regression modeling strategies with applications to linear models, logistic and ordinal regression, and survival analysis. Springer; 2015. — https://link.springer.com/book/10.1007/978-3-319-19425-7